CLINICAL TRIAL: NCT01018875
Title: A Randomized, Double-Blind, Active- and Placebo-Controlled Study to Evaluate the Efficacy and Safety of ABT-288 in Subjects With Mild-to-Moderate Alzheimer's Disease
Brief Title: Efficacy and Safety Study of ABT-288 in Subjects With Mild-to-Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-822; 2009-010704-29 (EudraCT Number)
Record Dates: First submitted 2009-11-20; First posted 2009-11-24 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2013-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-(4'-(5-methylhexahydropyrrolo(3,4-b)pyrrol-1-yl)biphenyl-4-yl)-2H-pyridazin-3-one; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1, Dose 1, ABT-288 (Experimental): Low Dose
  Interventions: Drug: ABT-288
- Arm 2, Dose 2, ABT-288 (Experimental): High dose
  Interventions: Drug: ABT-288
- donepezil (Active Comparator)
  Interventions: Drug: donepezil
- sugar pill (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ABT-288 — Subjects will take 4 capsules once daily for 12 weeks.
  Arms: Arm 1, Dose 1, ABT-288; Arm 2, Dose 2, ABT-288
Drug: donepezil — Subjects will take 4 capsules once daily for 12 weeks.
  Other Names: Aricept
  Arms: donepezil
Drug: placebo — Subjects will take 4 capsules once daily for 12 weeks.
  Arms: sugar pill

SUMMARY:
Efficacy and safety study of ABT-288 in adults with mild-to-moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria: 1. Have voluntarily signed an informed consent. 2. Subject meets diagnostic criteria criteria for probable AD (Alzheimer's Disease). 3. Female subjects must be postmenopausal for at least 2 years or surgically sterile. 4. Male subjects must be surgically sterile, sexually inactive or using a barrier method of birth control. 5. Subject has an identified, reliable caregiver. 6. Subject has a CT or MRI scan within 36 months prior to randomization. 7. With the exception of a diagnosis of mild-to-moderate AD and the presence of stable medical conditions, the subject is generally in good health based on medical history, physical examination, vital signs, clinical lab tests and ECG Exclusion Criteria: 1. Subject is currently taking or has taken a medication for the treatment of AD or dementia with 60 days of Screening visit, or is participating in cognitive therapy for the treatment of AD or dementia. 2. Subject uses non-prescribed drugs of abuse or has a history of drug or alcohol abuse/dependence. 3. Subject has a history of any significant neurologic disease other than AD. 4. Subject has a history of intolerance or adverse reaction to donepezil that led to discontinuation. 5. Subject has received any investigation product within 6 weeks prior to study drug administration.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
ADAS-cog: Alzheimer's Disease Assessment Scale - Cognition portion | Screening Visit 1 & 2, Day -1, Weeks 4, 8 & 12/PD

SECONDARY OUTCOMES:
MMSE: Mini Mental Status Exam | Screening Visit 1 & 2, Day -1, Weeks 4, 8 & 12/PD
NPI: Neuropsychiatric Inventory | Day -1, Weeks 4,8, 12/PD
ADCS-ADL: Alzheimer's Disease Cooperative Study | Day -1, Weeks 4,8 & 12/PD
CIBIC-Plus: Clinician Interview-Baed Impression of Change - plus | Day -1, Weeks 4,8 & 12/PD]

CONTACTS AND LOCATIONS:
Overall Officials: George Haig, Study Director — AbbVie
Locations (21):
- Russia (10):
  - Site Reference ID/Investigator# 22687, Kazan'
  - Site Reference ID/Investigator# 22636, Moscow
  - Site Reference ID/Investigator# 23702, Moscow
  - Site Reference ID/Investigator# 22635, Saint Petersburg
  - Site Reference ID/Investigator# 22633, Saint Petersburg
  - Site Reference ID/Investigator# 22637, Saint Petersburg
  - Site Reference ID/Investigator# 22632, Saint Petersburg
  - Site Reference ID/Investigator# 22634, Saint Petersburg
  - Site Reference ID/Investigator# 24563, Saint Petersburg
  - Site Reference ID/Investigator# 22689, Saratov
- Ukraine (11):
  - Site Reference ID/Investigator# 22630, Dnipro
  - Site Reference ID/Investigator# 22625, Donetsk
  - Site Reference ID/Investigator# 22624, Hlevakha
  - Site Reference ID/Investigator# 22629, Kharkiv
  - Site Reference ID/Investigator# 24565, Kherson
  - Site Reference ID/Investigator# 24566, Kiev
  - Site Reference ID/Investigator# 22622, Kiev
  - Site Reference ID/Investigator# 22623, Kiev
  - Site Reference ID/Investigator# 22628, Luhansk
  - Site Reference ID/Investigator# 43143, Odesa
  - Site Reference ID/Investigator# 22627, Poltava

REFERENCES:
- [Background] Hung SY, Fu WM. Drug candidates in clinical trials for Alzheimer's disease. J Biomed Sci. 2017 Jul 19;24(1):47. doi: 10.1186/s12929-017-0355-7. PMID 28720101